CLINICAL TRIAL: NCT06183086
Title: Prospective, Multicentre, Single-arm, Controlled Study on the Safety of Linovera® for the Treatment of Category-I Pressure Ulcers/Injuries
Brief Title: PMCF Study on the Safety of Linovera® for the Treatment of Category-I Pressure Ulcers/Injuries
Acronym: TRELINOIL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: B. Braun Medical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: BA-O-H-23029
Record Dates: First submitted 2023-10-19; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Linovera: Apply Linovera under clinical routine practice
  Interventions: Device: Linovera®

INTERVENTIONS:
Device: Linovera® — Apply Linovera® at least twice a day (recommended every 12 h) on the pressure ulcer/injury until Category-1 pressure ulcer/injury is healed or until discharge.

SUMMARY:
To assess the safety and performance of Linovera® in the treatment of Category- I pressure ulcers/injuries.

DETAILED DESCRIPTION:
The aim of this clinical study is to generate further clinical evidence for the use and benefit of Linovera® in the treatment of Category-I PUs. The results of this study will generate further clinical evidence for the use and the benefit of Linovera® in this indication.

Furthermore, the proactive collection of clinical data for Linovera® will support the maintenance of this skin oil on the market, so that in the future other patients can receive the product for the treatment of Category-I PUs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years)
* Patients with at least one Category-I PU/I (remark: follow-up will be done for one ulcer per patient).
* Provision of voluntary consent to participate in the study, following a full explanation of the nature and purpose of the study, by signing the informed consent form approved by the EC prior to all evaluations.
* Patient naïve to Linovera® 2 weeks before visit 1 (only applicable to the area of the skin that will be assessed).
* Patients which can be potentially followed until their Category-1 pressure ulcer/injury is healed throughout the duration of the study, according to the clinicians opinion.

Exclusion Criteria:

* Age <18 years
* Known allergies and/or hypersensitivity to any component of Linovera®.
* Any medical or psychological disorder that, in the investigator's opinion, may interfere with the patient's ability to give informed consent and comply with the study procedures.
* Any planned intervention that, in the investigator opinion, may affect skin condition of the patient (e.g. chemotherapy or radiotherapy).
* Simultaneous participation in an interventional clinical trial (drugs or medical devices studies).
* Any other additional topical treatments applied in the area of the skin that will be assessed.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See eligibility criteria
Sampling Method: Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Safety of Linovera® | From the date of start of study until Category-1 pressure ulcer/injury heals or patient discharge, whichever came first, assessed up to 30 days
  Number of patients with at least one Adverse Device Effect (ADE) or Severe Adverse Device Effect (SADE).

SECONDARY OUTCOMES:
Healing of the Category-1 pressure ulcer/injury | From the start of the study until the first 72 hours and when the Category-1 pressure ulcer/injury healed and/or at patient discharge
  Healing will be evaluated according to routine clinical practices with the following scale: Healed, no variation and worsening.
Patient and intended user satisfaction | From the start of the study until the first 72 hours and when the Category-1 pressure ulcer/injury healed and/or at patient discharge
  A Visual Analogue Scale will be used, 0 representing "very poor" and 100 representing "excellent".
Ease of use of the device | From the start of the study until Category-1 pressure ulcer/injury healed and/or at patient discharge, whichever came first, assessed up to 30 days
  The following paramenters will be evaluated by the patient and/or by the healthcare professional: ease of spreading surfaces, needed dose of oil dispensed, ease of application in large surfaces, absorption of Linovera®. This handling parameters will be rated as "very easy", "easy", "diffucult" or "very difficult".
Cumulative rates of each ADE/SADE | From the start of the study until Category-1 pressure ulcer/injury healed or patient discharge, whichever came first, assessed up to 30 days
  Cumulative rates of each ADE/SADE that might appear until the Category-1 pressure ulcer/injury has healed and/or until patient discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Susana Valerdiz, Principal Investigator — Hospital Universitario Central de Asturias
Locations (1):
- Hospital Universitario Central de Asturias, Oviedo, Spain

IPD SHARING:
Plan to Share IPD: Undecided